CLINICAL TRIAL: NCT02648581
Title: A Phase 2 Open-Label Study to Evaluate the Efficacy and Safety of Ustekinumab, a Human Monoclonal Anti-IL-12/IL-23 Antibody, in Patients With Behçet Disease
Brief Title: Efficacy and Safety of Ustekinumab, a Human Monoclonal Anti-IL-12/IL-23 Antibody, in Patients With Behçet Disease
Acronym: STELABEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P140302
Record Dates: First submitted 2015-12-21; First posted 2016-01-07 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Behçet Disease
Keywords: Behçet; ulcers; uveitis; ustekinumab; biologics
MeSH Terms: conditions — Behcet Syndrome; Ulcer; Uveitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subcutaneous Ustekinumab (Experimental)
  Interventions: Drug: Subcutaneous Ustekinumab

INTERVENTIONS:
Drug: Subcutaneous Ustekinumab — Injections of ustekinumab at 90 mg at week 0, week 4 and week 16. Patients in treatment failure at week 24 will terminate the study. Responder patients at week 24 will receive additional 2 injections of ustekinumab at week 28 and week 40 with a final evaluation at week 52.

SUMMARY:
The purpose of this study is to evaluate the proof of concept of efficacy of ustekinumab in subjects with Behçet disease, including patients with oral ulcers (STELABEC-1) and patients with active posterior uveitis or panuveitis (STELABEC-2)

DETAILED DESCRIPTION:
Behçet disease (BD) is a chronic systemic inflammatory disorder at the crossroad between autoimmune and autoinflammatory syndromes. Two recent large genome-wide association studies (GWAS) conducted in Turkey and Japan reported association between single nucleotide polymorphism (SNP) of interleukin (IL)-10 and IL-23R/IL-12RB2 genes and BD. Interleukin-12 and interleukin-23, cytokines that induce naive CD4+ lymphocytes to differentiate into type 1 helper T cells (Th1 cells) and type 17 helper T cells (Th17 cells), respectively, have been identified as key mediators of BD. Promotion of Th1 and Th17 responses and suppression of regulatory T cells correlate with BD activity.

Due to the lack of an etiologic agent, the treatment is symptomatic without consensus. The goals are the functional recovery of a visceral involvement (eye, central nervous system) and prevention of relapse(s). The risks of BD are an increased mortality especially in case of arterial involvement, and a high morbidity due to the cumulative sequelae of ocular and neurological involvement. Steroids are the corner stone of the antiinflammatory agents administered topically or systemically. Relapses are frequently seen after discontinuation of steroids, and corticodependence is frequently observed leading to the use of immunosuppressive drugs.

Biologic agents that selectively block steps in the inflammatory cascade could provide additional therapies for BD.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age.
2. Have a diagnosis of BD according to the International Classification Criteria (criteria from the International Study Group and/or the 2013 International Criteria for BD).
3. Have an active disease at screening, defined by the presence of :

   For the STELABEC-1 study : Recurrent oral and/or genital ulcers, defined as ≥2 episodes within 3 months before study entry. Before study entry, patients should have at least 2 oral ulcers within the last 2 weeks before baseline visit.

   For the STELABEC-2 study : Active posterior uveitis and/or panuveitis and/or retinal vasculitis, defined by the presence of at least 1 or the following parameters in at least one eye :
   * Active, inflammatory, chorioretinal and/or inflammatory retinal vascular lesion
   * ≥2+ anterior chamber cells (Standardization of Uveitis Nomenclature [SUN] criteria)
   * ≥2+ vitreous haze (National Eye Institute [NEI]/SUN criteria)
4. Have previously received at least 1 non-biologic therapy :

   For the STELABEC-1 study : Colchicine ≥1 mg/day for all patients For the STELABEC-2 study : Subjects must have active disease at the baseline visit despite at least 2 weeks of oral prednisone ≥ 10 mg/day to ≤60 mg/day (or oral corticosteroid equivalent) with or without prior high dose corticoid pulse.
5. Are without treatment regimen (due to ineffectiveness / intolerance) or on a stable BC treatment regimen consisting of any of the following medications (alone or in combination) : Corticosteroids for a period of at least 2 weeks prior to Day 0 Colchicine for a period of at least 30 days prior to Day 0 Immunosuppressive or immunomodulatory agents for a period of at least 30 days prior to Day 0 Thalidomide for a period of at least 60 days prior to Day 0
6. A female subject is eligible to enter the study if she is :

   * Not pregnant or breast-feeding
   * Of non-childbearing potential (ie, women who had a hysterectomy, are postmenopausal which is defined as 1 year without menses, have both ovaries surgically removed or have current documented tubal ligation); or
   * Of childbearing potential (ie, women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea [even severe], women who are perimenopausal or have just begun to menstruate. These women must have a negative serum pregnancy test at screening, and agree to 1 of the following :

   Complete abstinence from intercourse from 2 weeks prior to administration of the 1st dose of study agent until 8 weeks after the last dose of study agent; or

   Consistent and correct use of 1 of the following acceptable methods of birth control for 1 month prior to the start of the study agent and 15 weeks after the last dose of study agent :
   * Implants of levonorgestrel;
   * Injectable progesterone;
   * Any intrauterine device (IUD) with a documented failure rate of less than 1% per year;
   * Oral contraceptives (either combined or progesterone only);
   * Double barrier method: Condom, cervical cap or diaphragm with spermicidal agent;
   * Transdermal contraceptive patch;
   * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for the female subject.
7. Have the ability to understand the requirements of the study provide written informed consent (including consent for the use and disclosure of research-related health information) and comply with the study protocol procedures (including required study visits).
8. Affiliation with a mode of social security (profit or being entitled)

Exclusion Criteria:

* Have required 3 or more courses of systemic corticosteroids for concomitant conditions (eg, asthma, atopic dermatitis) within 90 days of Day 0 (Topical or inhaled steroids are permitted)
* Have received intravenous (IV) or oral cyclophosphamide within 180 days of Day 0.
* Have received any of the following within 90 days of Day 0 :

Anti-TNF therapy (eg, adalimumab, etanercept, infliximab). Interleukin-1 receptor antagonist (anakinra). Abatacept Interleukin-6 receptor antagonist (tocilizumab) Intravenous immunoglobulin (IVIG) High dose prednisone (> 100 mg/day).

* Have received any of the following within 60 days of Day 0 :

A non-biologic investigational agent. Any new immunosuppressive/immunomodulatory agent. Any steroid injection (intramuscular, intraarticular or intravenous).

* Have received any of the following within 30 days of Day 0 :

A live vaccine within 30 days of Day 0. A change in dose of a corticosteroid within 2 weeks days of Day 0. A change in dose of other immunosuppressive/immunomodulatory agent within 30 days of Day 0.

* Have very severe Behçet disease (defined by current severe complication of BD: digestive, cardiac, pulmonary or central nervous system involvement assessed as very severe by the referring clinician) requiring high dose prednisone (≥1mg/kg) within 30 days of Day 0 (with the exception of high dose prednisone pulse for active uveitis)
* Have a history of a major organ transplant (eg, heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to BD which, in the opinion of the principal investigator, could confound the results of the study or put the subject at undue risk.
* Have a planned surgical procedure or a history of any other.
* Medical disease, laboratory abnormality, or condition that, in the opinion of the principal investigator, makes the subject unsuitable for the study.
* Have a history of malignant neoplasm within the last 5 years, except for treated cancers of the skin or carcinoma in situ of the uterine cervix.
* Have required management of acute or chronic infections :

  * Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria).
  * Hospitalization for treatment of infection within 60 days of Day 0.
  * Use of parenteral (IV or IM) antibiotics (antibacterials, antivirals, anti-fungals, or anti parasitic agents) within 60 days of Day 0.
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Day 0.
* Have a historically positive test or test positive at screening for HIV-1 antibody, hepatitis C virus antibodies, hepatitis B surface antigen (HbsAg), or antiHBcAg positivity (without HbsAg positivity).
* Have a Grade 3 or greater laboratory abnormality based on the protocol toxicity scale except for the following that are allowed:

  * Stable Grade 3 prothrombin time (PT) secondary to warfarin treatment.
  * Stable Grade 3/4 proteinuria (≤ 6 g/24 hour equivalent by spot urine protein to creatinine ratio allowed).
  * Stable Grade 3 neutropenia or stable Grade 3 white blood cell count.
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Number of oral ulcers at week 24 compared to baseline | 24 weeks
  Treatment efficacy at week 24 for STELABEC-1 study on oral ulcers
Number of uveitis or retinal vasculitis remission | 24 weeks
  Treatment efficacy at week 24 for STELABEC-2 study on eye involvement

SECONDARY OUTCOMES:
Number of oral and genital ulcers | at baseline visit (week 0)
Number of oral and genital ulcers | 4 weeks
Number of oral and genital ulcers | 8 weeks
Number of oral and genital ulcers | 12 weeks
Number of oral and genital ulcers | 16 weeks
Number of oral and genital ulcers | 24 weeks
Number of oral and genital ulcers | 28 weeks
Number of oral and genital ulcers | 40 weeks
Number of oral and genital ulcers | 52 weeks
Pain Visual Analog Scales of oral and genital ulcers | at baseline visit (week 0)
Pain Visual Analog Scales of oral and genital ulcers | 4 weeks
Pain Visual Analog Scales of oral and genital ulcers | 8 weeks
Pain Visual Analog Scales of oral and genital ulcers | 12 weeks
Pain Visual Analog Scales of oral and genital ulcers | 16weeks
Pain Visual Analog Scales of oral and genital ulcers | 24 weeks
Pain Visual Analog Scales of oral and genital ulcers | 28 weeks
Pain Visual Analog Scales of oral and genital ulcers | 40 weeks
Pain Visual Analog Scales of oral and genital ulcers | 52 weeks
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | baseline visit (week 0)
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | 4 weeks
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | 8 weeks
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | 12 weeks
Visual acuity by Early Treatment Diabetic Retinopathy Study (ETDRS) | 16 weeks
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | 24 weeks
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | 28 weeks
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | 40 weeks
Number of chorioretinal and/or inflammatory retinal vascular lesions, inflammation in anterior chamber and in vitreous haze | 52 weeks
Behçet Syndrome Activity Score (BSAS) | 12 weeks
Behçet Disease Current Activity Form (BDCAF) | 12 weeks
Behçet Syndrome Activity Score (BSAS) | 24 weeks
Behçet Disease Current Activity Form (BDCAF) | 24 weeks
Behçet Syndrome Activity Score (BSAS) | 52 weeks
Behçet Disease Current Activity Form (BDCAF) | 52 weeks
Behçet Disease Quality of Life Measure : Short Form-36 (SF- 36) | 12 weeks
Behçet Disease Quality of Life Measure : Routine Assessment of Patient Index Data 3 (RAPID3) | 12 weeks
Behçet Disease Quality of Life Measure : Short Form-36 (SF- 36) | 24 weeks
Behçet Disease Quality of Life Measure : Routine Assessment of Patient Index Data 3 (RAPID3) | 24 weeks
Behçet Disease Quality of Life Measure : Short Form-36 (SF- 36) | 52 weeks
Behçet Disease Quality of Life Measure : Routine Assessment of Patient Index Data 3 (RAPID3) | 52 weeks
Number of adverse events | from baseline visit up to 52 weeks
  adverse events including headache, arthralgia, infection (pneumonia and bronchitis),skin infections, shingles, depression, dizziness, diarrhea, pruritus, myalgia, asthenia

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin TERRIER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Department of Internal Medicine, National Reference Center for Autoimmune and Systemic Diseases, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Revel MP, Chassagnon G, Sanchez O, Ferretti G, Millet I, Rocher L, Maitre S, Lederlin M, Ducou-le-Pointe H, Rousset P, Bennani S, Zins M, Bruneau B, Tissot V, Alison M, Canniff E, Siauve N, Vandeventer S, Le Blanche AF, Planquette B, Tsatsaris V, Coste J. CT venography for the diagnosis of postpartum venous thromboembolism: a prospective multi-center cohort study. Eur Radiol. 2024 Nov;34(11):7419-7428. doi: 10.1007/s00330-024-10791-8. Epub 2024 May 23. PMID 38782788
- [Background] London J, Regent A, Dion J, Jilet L, Jachiet M, Lidove O, Cohen-Aubart F, Aractingi S, Guegan S, Pennaforte JL, Abdoul H, Puechal X, Terrier B. Efficacy and safety of ustekinumab in Behcet disease: Results from the prospective phase 2 STELABEC trial. J Am Acad Dermatol. 2022 Sep;87(3):681-684. doi: 10.1016/j.jaad.2021.11.045. Epub 2021 Dec 2. No abstract available. PMID 34864108